CLINICAL TRIAL: NCT02058914
Title: Moderate Amounts of High Fructose- or High Glucose-sweetened Beverages do Not Differentially Alter Metabolic Health in Male and Female Adolescents
Brief Title: Effects of Sugar Sweetened Beverage on Metabolic Health in Male and Female Adolescents
Acronym: adol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: fructadol
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Insulin Sensitivity; Insulin Tolerance
Keywords: Sugar sweetened beverages; metabolism; endocrine; lipids; blood glucose
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high fructose sweetened beverage (Experimental): 710 ml per day of a HF-sweetened beverage (sweetened with 50 g fructose and 15 g glucose)
  Interventions: Dietary Supplement: high fructose sweetened beverage
- High Glucose sweetened beverage (Active Comparator): HG-sweetened beverage (sweetened with 50 g glucose and 15 g fructose)
  Interventions: Dietary Supplement: High Glucose sweetened beverage

INTERVENTIONS:
Dietary Supplement: high fructose sweetened beverage — 710 ml per day of a HF-sweetened beverage
  Arms: high fructose sweetened beverage
Dietary Supplement: High Glucose sweetened beverage — HG-sweetened beverage
  Arms: High Glucose sweetened beverage

SUMMARY:
We examined the effects of short-term (2-wk) consumption of HF- and HG-sweetened beverages in adolescents (15-20 yr of age) on insulin sensitivity, insulin secretion, insulin clearance, triacylglycerol (TAG), and cholesterol concentrations.

DETAILED DESCRIPTION:
This counterbalanced study consisted of two trials including 1) high fructose (HF) trial and, 2) a high glucose (HG) trial. Each trial was blind to the participant, performed in a random order, and was 15 d in length. During days 1-14 of each trial, the participants consumed either 710 ml per day of a HF-sweetened beverage (sweetened with 50 g fructose and 15 g glucose) for 2-wk (HF trial) or 710 ml per day of a HG-sweetened beverage (sweetened with 50 g glucose and 15 g fructose) for 2-wk (HG trial) on top of their normal diet. In addition, the participants were instructed to maintain their normal physical activity levels during each trial (which were measured with an accelerometer). On day 15 of each trial, the participants reported to the lab after a ~ 11 h overnight fast for metabolic testing. During this testing day, the participants remained in the lab for 12 h and consumed three liquid meals (one meal every 4 h and HF meals during HF trial and HG meals during HG trial), while blood samples were taken every 15 or 30 min throughout the 12 h testing day. During testing, the participants remained physically inactive (< 3,000 steps).

ELIGIBILITY:
Inclusion Criteria:

males and females 15-20 years of age not participating in an organized sport (non-athletes) no history of heart, lung, kidney, endocrine, or gastrointestinal disease no medications known to alter glucose or lipid metabolism normal fasting blood glucose concentrations (< 100 mg/dL) normal fasting triglyceride concentrations (< 150 mg/dL) average daily fructose consumption < 90th percentile for age and sex

Exclusion Criteria:

athlete type 1 diabetic type 2 diabetic consuming high quantities of fructose

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
glucose concentrations | baseline and 15, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 255, 270, 285, 300, 315, 330, 360, 390, 420, 450, 480, 495, 510, 525, 540, 555, 570, 600, 630, 660, 690, and 720

SECONDARY OUTCOMES:
Triglycerides | baseline and 15, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 255, 270, 285, 300, 315, 330, 360, 390, 420, 450, 480, 495, 510, 525, 540, 555, 570, 600, 630, 660, 690, and 720

OTHER OUTCOMES:
insulin | baseline and 15, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 255, 270, 285, 300, 315, 330, 360, 390, 420, 450, 480, 495, 510, 525, 540, 555, 570, 600, 630, 660, 690, and 720

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heden TD, Liu Y, Park YM, Nyhoff LM, Winn NC, Kanaley JA. Moderate amounts of fructose- or glucose-sweetened beverages do not differentially alter metabolic health in male and female adolescents. Am J Clin Nutr. 2014 Sep;100(3):796-805. doi: 10.3945/ajcn.113.081232. Epub 2014 Jul 16. PMID 25030782